CLINICAL TRIAL: NCT06850298
Title: Investigation of Impact of Milk Consumption on H5 Influenza Detection in Respiratory Specimens
Brief Title: H5N1 Milk Detection Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Daniel S. Graciaa, MD, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009067; 75N93021C00017-P00012-9999-5 (NIH)
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Influenza
Keywords: Pasteurized Milk; Flu Virus A (H5); H5N1 avian influenza A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1-Day Group (Experimental): Participants will consume 250 mL of pasteurized commercial milk at a study visit.
  Interventions: Other: Pasteurized milk contaminated with killed A(H5) virus
- 3-Day Group (Experimental): Participants will consume 250 mL of pasteurized commercial milk for a total of 3 daily consecutive visits.
  Interventions: Other: Pasteurized milk contaminated with killed A(H5) virus

INTERVENTIONS:
Other: Pasteurized milk contaminated with killed A(H5) virus — Milk to be used in the study will be obtained from the CDC. Pasteurized commercial milk likely to contain detectable A(H5N1) particles will be obtained from a source such as a recently affected dairy farm. The CDC Influenza Division laboratory (Viral, Surveillance, and Diagnosis Branch) will test the milk to confirm the presence of viral A(H5) RNA using a protocol developed and validated by the US FDA Agricultural Research Service. The US Food and Drug Administration (FDA) has indicated that the consumption of commercial pasteurized dairy products in the US is safe.

SUMMARY:
The purpose of this study is to determine whether drinking pasteurized milk (milk heated to kill harmful germs) that contains inactive particles of a flu virus called A(H5) could lead to the detection of the virus in the nose or throat. Inactive particles are not capable of causing disease. The results will help the Centers for Disease Control and Prevention (CDC) better understand how milk consumption could affect flu surveillance. Investigators also want to see if the body produces antibodies in response to this milk consumption.

DETAILED DESCRIPTION:
Since March 2024, avian influenza A (H5N1) viruses have infected U.S. dairy cattle and spread widely. The virus has been identified in high concentrations in raw milk, and research shows that pasteurization - the process of heating milk to a specific temperature for a set time - inactivates the A (H5N1) virus. Therefore, the Food and Drug Administration (FDA) says that commercial pasteurized milk is safe for consumption. However, trace amounts of inactive influenza particles may still be detected in pasteurized milk.

This study aims to determine whether drinking pasteurized milk could be a possible exposure for H5N1 influenza detection. The findings will support the Centers for Disease Control and Prevention's (CDC) efforts to evaluate milk consumption as a factor in influenza surveillance and provide context for interpreting surveillance data.

Healthy adults will drink 250 mL of pasteurized milk containing the inactive H5N1 virus, provided by the CDC, either during a single visit or over three consecutive daily visits. Nasal and combined nasal/oral swabs will be collected immediately following milk consumption to assess the presence of influenza. Additionally, a subset of participants will provide blood, saliva, and stool samples at the initial visit and again 21-30 days post-consumption.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-64 years
* BMI ≤ 35 kg/m2
* Able to understand and give informed consent (American English) and comply with study visits and procedures.
* In good general health based on medical history and the investigator's clinical judgment.

Exclusion Criteria:

* Symptoms of acute respiratory illness or conjunctivitis within 7 days
* Febrile illness in the previous 72 hours
* Recent influenza antiviral use (within 14 days)
* Immunosuppression due to illness or medications
* Current pregnancy or breastfeeding
* History of allergy or intolerance to milk or milk alternatives
* Consumption of raw (unpasteurized) milk within the previous 14 days
* Recent work (within 14 days) on a farm with animals known to be infected with A(H5) virus
* Previous receipt of A(H5) vaccine at any time

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of respiratory specimens with influenza detected | Up to 30 days after milk consumption
  Proportion of respiratory specimens (nasopharyngeal and combined nasal/oropharyngeal swabs) with detection of influenza after consumption of pasteurized milk contaminated with killed A(H5) virus

SECONDARY OUTCOMES:
Severe adverse events after milk consumption | Up to 30 days after milk consumption
  Participants will be asked to call the site if they develop any adverse events for the entire the study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Graciaa, MD, MPH, MSc, Principal Investigator — Emory University
Locations (1):
- Hope Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share deidentified respiratory testing results.
Supporting Information: Study Protocol
Time Frame: The team will share the data immediately following the study publication, or at the end of the study analysis if not published, with no end date.
Access Criteria: Data will be available for access in a public database such as Dataverse.